CLINICAL TRIAL: NCT05883397
Title: Enhanced Hippocampal Neuroplasticity for Surfacing of Inaccessible Traumatic Memories in Veterans With PTSD
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Collaborators: Weizmann Institute of Science (Other); Office of Naval Research (ONR) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 90-22
Record Dates: First submitted 2023-03-05; First posted 2023-06-01 (Actual); Last update posted 2023-06-01 (Actual); Status verified 2023-05

CONDITIONS: PTSD; Peritraumatic Amnesia
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be recruited from veterans' clinics and veterans' organizations. After screening, eligible participants will undergo baseline evaluation. Enrolled participants will be 1:1 randomly assigned to the HBOT or HBOT + hippocampal training, according to a computer-generated randomization list. Assessors will be blinded to the participants' allocation.
  During the study period, all the participants will continue their psychological and pharmacological treatment as prior to their inclusion in the study. Any changes in the frequency of psychologic treatment or pharmacotherapy dose will be reported and documented.
  The study is designed as a per protocol trial, and thus, participants will only be included in the analysis if they completed the treatment protocol and attained study analysis.
Who Masked: Care Provider, Investigator, Outcomes Assessor
Masking Description: Care providers, Investigator and assessors will be blinded to the participants' allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HBOT (Active Comparator): Participants will be treated in a multiplace chamber (HAUX-Life-Support GmbH) for a total of 60 daily sessions, five days a week. Each session will consist of 90 minutes exposure to 100% oxygen at 2 ATA (atmospheres), with five-minute air brakes every 20 minutes.
  Interventions: Other: HBOT
- HBOT + hippocampal training (Active Comparator): Participants will be treated in a multiplace chamber (HAUX-Life-Support GmbH) for a total of 60 daily sessions, five days a week. Each session will consist of 90 minutes exposure to 100% oxygen at 2 ATA, with five-minute air breaks every 20 minutes.
  Hippocampal training: This will combine physical and cognitive training. Training will be given 3 times per week, prior to the next HBOT, and more than 20 hours after the last HBOT session.
  Interventions: Other: HBOT; Other: Hippocampal training

INTERVENTIONS:
Other: HBOT — Participants will be treated in a multiplace chamber (HAUX-Life-Support GmbH) for a total of 60 daily sessions, five days a week. Each session will consist of 90 minutes exposure to 100% oxygen at 2 ATA, with five-minute air breaks every 20 minutes.
Other: Hippocampal training — Hippocampal training: This will combine physical and cognitive training. Training will be given 3 times per week, prior to the next HBOT, and more than 20 hours after the last HBOT session.
  Arms: HBOT + hippocampal training

SUMMARY:
Hyperbaric oxygen therapy (HBOT) includes the inhalation of 100% oxygen at pressures exceeding one atmosphere absolute. HBOT has been applied worldwide, mostly for chronic non-healing wounds. Our team demonstrated that HBOT induced hippocampal neuroplasticity in veterans with long-standing treatment-resistant PTSD; this led to enhanced memory recovery and significant improvement in PTSD symptoms.

Both physical activity, such as aerobic exercise, and cognitive training were shown to support neurogenesis in the hippocampus. Therefore, the current study aims to evaluate whether hippocampal training, induced by physical and cognitive training, will augment the hippocampal neuroplasticity effect of HBOT and further enhance recovery of inaccessible memories in veterans with PTSD.

The protocol will include forty male veterans aged 25 to 60 years, with combat-associated PTSD and peritraumatic amnesia, who will receive either HBOT alone or HBOT and hippocampal training. The HBOT protocol will consist of 60 daily sessions, 90-minutes each, five days a week. Hippocampal training will combine physical and cognitive training 3 times per week, prior to HBOT sessions. Detailed psychological evaluation, anatomic and functional MRI, electroencephalogram and autonomic nervous system data will be obtained at baseline, and during and after treatment.

The proposed study offers a new approach of biological treatment for memory manipulations. The findings will help elucidate the mechanism of PTSD-related memory impairment and is expected to contribute to the development of biological memory manipulations for treating PTSD and other memory-related conditions.

DETAILED DESCRIPTION:
Our memory constructs a sense of coherence and defines the way we perceive the world. Effective encoding of memories in an adequate context, and their deliberate retrieval at a later time, are crucial for maintaining biographic continuity, and are both heavily dependent on hippocampal function.

Post-traumatic stress disorder (PTSD) can be considered a prototype disorder in which a stressogenic event leads to hippocampal malfunction and mal-encoding of a traumatic memory. Persistent hippocampal dysfunction contributes to the unremitting nature of PTSD years after the acute event. The upshot is not only amnesia, but also difficulty in memory integration in the context of time and location, and the feeling that the traumatic event is present all the time and everywhere. Improved hippocampal function may contribute to better access to memories of a traumatic event and to memory contextualization and neutralization. Memory processing is essential for PTSD recovery.

Hyperbaric oxygen therapy (HBOT) includes the inhalation of 100% oxygen at pressures exceeding one atmosphere absolute. HBOT has been applied worldwide, mostly for chronic non-healing wounds. Our team demonstrated that HBOT induced hippocampal neuroplasticity in veterans with long-standing treatment-resistant PTSD; this led to enhanced memory recovery and significant improvement in PTSD symptoms. The investigators also demonstrated effects of HBOT on memory recovery among women with fibromyalgia due to childhood sexual abuse.

Both physical activity, such as aerobic exercise, and cognitive training were shown to support neurogenesis in the hippocampus. Therefore, the current study aims to evaluate whether hippocampal training, induced by physical and cognitive training, will augment the hippocampal neuroplasticity effect of HBOT and further enhance recovery of inaccessible memories in veterans with PTSD.

The protocol will include forty male veterans aged 25 to 60 years, with combat-associated PTSD and peritraumatic amnesia, who will receive either HBOT alone or HBOT and hippocampal training. The HBOT protocol will consist of 60 daily sessions, 90-minutes each, five days a week. Hippocampal training will combine physical and cognitive training 3 times per week, prior to HBOT sessions. Detailed psychological evaluation, anatomic and functional MRI, electroencephalogram and autonomic nervous system data will be obtained at baseline, and during and after treatment.

The proposed study offers a new approach of biological treatment for memory manipulations. The findings will help elucidate the mechanism of PTSD-related memory impairment, and is expected to contribute to the development of biological memory manipulations for treating PTSD and other memory-related conditions.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of PTSD
* A history of trauma of at least one course of trauma-focused psychotherapy
* The presence of peri-traumatic amnesia

Exclusion Criteria:

* A history of traumatic brain injury or any other known brain pathology except PTSD
* Active smoking
* Drugs or alcohol abuse other than prescribed cannabis
* Active asthma, lung pathology, epilepsy or otolaryngological disease incompatible with HBOT
* The presence of shards or another contraindication for MRI

Ages: 25 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Only male will be recruited to the study
Enrollment: 60 (Estimated)
Dates: Start 2023-05-25 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Changes in memory gaps (as assessed by the traumatic scene form) | through study completion, an average of 4 months
  traumatic scene form will be used to assess memory gaps. The intensity of each part sensation will be scored between 0 and 10 (higher score reflects stronger memory). A time line of the event will be drown, and amnestic parts of the memory will be marked (the presumed amnestic time will be evaluated in minutes)
Time to inaccessible memory surfacing | through study completion, an average of 4 months
  Daily questionnaire will be used to assess surfacing of new memories. The time of memory surfacing will be defined (session number)

SECONDARY OUTCOMES:
Change in brain activity as assessed by fMRI (functional magnetic resonance imaging) | through study completion, an average of 4 months
  Three different fMRI paradigms will be used to assess hippocampal function, prefrontal cortex activity and the response to the traumatic memory
cognitive performance as assessed using "Neurotrax" | through study completion, an average of 4 months
  Global Score is calculated based on the scores given for Memory performance, Attention, Information Processing speed, Executive Function and Motor skills.
  The score ranges between 0 and 100, and higher score reflects better performance.
RAVLT memory test | through study completion, an average of 4 months
  The test is designed as a list-learning paradigm in which the patient hears a list of 15 nouns and is asked to recall as many words from the list as possible. After five repetitions of free-recall, a second "interference" list (List B) is presented in the same manner, and the participant is asked to recall as many words from List B as possible. After the interference trial, the participant is immediately asked to recall the words from List A, which she or he heard five times previously. After a 20 min delay, the participant is asked to again recall the words from List A. After this "delayed recall" task, a list of 50 words is presented containing all of the words from Lists A and B, in addition to 20 phonemically and/or semantically similar words. The multiple memory processes assessed as a global score, called "Total Learning" The score ranges between 0 and 100, and higher score reflects better performance.
ROCFT memory test | through study completion, an average of 4 months
  Copy Z Immediate recall Raw Delayed recall Z will be used to evaluate memory performance, higher scores reflects better performance.
Verbal Pairs memory test | through study completion, an average of 4 months
  Recall Total Score First Recall Total Score Learning Slope Delayed List Recall Score Percent retention Recognition Score will be used to evaluate memory performance, higher scores reflects better performance.

CONTACTS AND LOCATIONS:
Locations (1):
- Assaf-Harofeh Medical Center, Ramla, Israel

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared with other researches.